CLINICAL TRIAL: NCT06490614
Title: Comparative Study Between Dexmedetomidine and Nalbuphine as Analgesic Adjuvants to Bupivacaine in Superficial Cervical Block for Patients Undergoing Anterior Cervical Discectomy and Fusion (ACDF) Surgery A Double Blinded Randomized Trial
Brief Title: Dexmedetomidine and Nalbuphine as Analgesic Adjuvants to Bupivacaine in Superficial Cervical Block.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Doaa Fawzy Abd El Fattah Hassan, Lecturer of anesthesia,surgical ICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-568-2023
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cervical Discectomy and Fusion (ACDF)
MeSH Terms: interventions — Dexmedetomidine; Nalbuphine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups in parallel for the duration of the study, either group A (Dexmedetomidine group) or group B (nalbuphine group).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will be subjected to SCPB consisting of bupivacaine 0.25%, dexmedetomidine 1 μg/kg (precedex 100mcg/ml), and adrenaline 1:200,000 in a total volume of 10ml normal saline.
  Interventions: Drug: Dexmedetomidine in superficial cervical plexus block
- Nalbuphine group (Experimental): Patients will be subjected to SCPB consisting of bupivacaine 0.25% and 10 mg of Nalbuphine (nalufin 20mg/ml) and adrenaline 1:200,000 in a total volume of 10ml normal saline.
  Interventions: Drug: Nalbuphine in superficial cervical plexus block

INTERVENTIONS:
Drug: Dexmedetomidine in superficial cervical plexus block — While the patient is in the supine position, the head will be turned to the opposite side of the surgical incision, and a line extending from the mastoid process to the clavicular head of the sternomastoid muscle will be marked. Aseptic preparation of this area will be done, and then the block needle will be inserted at the midpoint of this line with injection of bupivacaine 0.25%, dexmedetomidine 1 μg/kg (precedex 100mcg/ml), and adrenaline 1:200,000 in a total volume of 10ml normal saline in the above, below, and middle directions subcutaneously, creating a sausage-shaped swelling. The sensory block will be assessed with ice chips in the dermatome corresponding to the block, which included the skin of the neck, upper chest, shoulder, and ear, until the completion of the sensory blockade.
  Other Names: Percedex
  Arms: Dexmedetomidine group
Drug: Nalbuphine in superficial cervical plexus block — While the patient is in the supine position, the head will be turned to the opposite side of the surgical incision, and a line extending from the mastoid process to the clavicular head of the sternomastoid muscle will be marked. Aseptic preparation of this area will be done, and then the block needle will be inserted at the midpoint of this line with injection of bupivacaine 0.25%, 10 mg of Nalbuphine (nalufin 20mg/ml), and adrenaline 1:200,000 in a total volume of 10ml normal saline in the above, below, and middle directions subcutaneously, creating a sausage-shaped swelling. The sensory block will be assessed with ice chips in the dermatome corresponding to the block, which included the skin of the neck, upper chest, shoulder, and ear, until the completion of the sensory blockade.
  Other Names: Nalufin
  Arms: Nalbuphine group

SUMMARY:
Anterior cervical discectomy and fusion (ACDF) nowadays is considered a common procedure.postoperative pain can hinder recovery and prolong hospital stay. The superficial cervical plexus block (SCPB) is a safe and simple technique that had been found to allow good pain relief in neck surgeries. The main drawback of SCPB was short duration, so adjuvants as dexmedetomidine and opioids has been used to increase analgesic duration and decrease the use of opioids.

The current study will compare the efficacy of dexmedetomidine and nalbuphine as adjuvants to bupivacaine in SCPB in anterior cervical fusion surgeries.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate whether the addition of Dexmedetomidine to bupivacaine is comparable to the addition of nalbuphine in superficial cervical plexus block in patients undergoing ACDF.

thrity patients will be recruited. Patients will be divided randomly into either group A in which patients will receive SCPB consisting of bupivacaine 0.25%, dexmedetomidine 1 μg/kg (precedex 100mcg/ml), and adrenaline 1:200,000 in a total volume of 10ml normal saline, or Group B in which patients will receive SCPB consisting of bupivacaine 0.25% and 10 mg of Nalbuphine (nalufin 20mg/ml) and adrenaline 1:200,000 in a total volume of 10ml normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA I and ASA ll.
* Both males and females
* Age 21- 60 years.
* Patients undergoing elective anterior cervical discectomy and fusion for 1 or 2 levels.

Exclusion Criteria:

* Patient refusal.
* Patients undergoing anterior cervical vertebrectomy and reconstruction.
* Patients with a history of allergy to local anesthetics or any used drugs in study.
* Infection at the site of the block.
* Patients with multiple cervical spine traumas.
* Patients having surgery for malignant tumors.
* Pre-existing peripheral neuropathies.
* Pregnant female.
* Patients with uncontrolled hypertension or cardiac problems as (heart block, sick sinus syndrome and ischemic heart disease).
* Patients with coagulopathy (INR>1.5).
* Patients with failed block.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The total nalbuphine consumption in mg | The 1st 48 hours starting after patient transfer to the PACU.
  The total nalbuphine consumption measured in mg during the 1st 48 hours postoperatively starting after patient transfer to the PACU.

SECONDARY OUTCOMES:
Postoperative visual analogue scale (VAS) pain score | At 2, 4, 8, 12, 18, and 24 ,36 and 48 hours postoperatively .
  Postoperative ( visual analogue scale)VAS pain score , It consists of a 10 cm line with two anchor points zero means'no pain' and 10 is the worst pain imaginable' which is self-assessed by patients.
  VAS will be assessed at 2, 4, 8, 12, 18, and 24 ,36 and 48 hours
Time to first postoperative rescue analgesia | Postoperative 48 hours
  Time to first postoperative rescue analgesia(nalbuphine in incremental doses of 0.1 mg/kg and not exceeding 0.4 mg/kg in 2 hours) in hours.
heart rate (beats/min) | At baseline, every half an hour intraoperatively and at 2, 4, 8, 12, 18, 36, and 48 hours postoperatively.
  Intraoperative and postoperative heart rate HR (beats/min) in the two groups will be recorded at baseline, every half an hour intraoperatively and at 2, 4, 8, 12, 18, 36, and 48 hours postoperatively.
Ramsay Sedation Scale | 30 min, 1, 2, 4, 6, and 12, 36 and 48 hours postoperatively.
  Ramsay Sedation Scale , which divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. It will be measured at 30 min, 1, 2, 4, 6, and 12, 36 and 48 hours
  Ramsay sedation score:
  Awake level
  1. Anxious and agitated or restless, or both.
  2. Co-operative, oriented, and tranquil.
  3. Responds to commands only. Asleep level
  4. Brisk response to light glabellar tap or loud auditory stimulus.
  5. Sluggish response to light glabellar tap or loud auditory stimulus.
  6. Exhibits no response
Incidence of postoperative complications | Postoperative 48 hours
  Incidence of hypotension (MAP< 25% of baseline), bradycardia (HR< 50 bpm), respiratory rate < 10/min or postoperative nausea and vomiting
Mean arterial blood pressure (MAP) | Intraoperatively ,at baseline and every half an hour till the end of surgery, then at 2,4,8,12,18,36 and 48 hours postoperatively.
  Mean arterial blood pressure will be recorded intraoperatively and postoperatively at baseline and every half an hour till the end of surgery, then at 2, 4, 8,12,18, 36 and 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa F El Hamalawy, Lecturer, Study Director — Kasr Al-Aini hospital-Faculty of Medicine- Cairo University

REFERENCES:
- [Background] Rostami M, Moghadam N, Obeid I, Jouibari MF, Zarei M, Moosavi M, Khoshnevisan A, Farahbakhsh F, Moosaie F, Ehteshami S, Borghei A, Shafizadeh M, Kordi R, Khadivi M. The Impact of Single-Level Anterior Cervical Discectomy and Fusion on Cervical Sagittal Parameters and Its Correlation With Pain and Functional Outcome of Patients With Neck Pain. Int J Spine Surg. 2021 Oct;15(5):899-905. doi: 10.14444/8115. Epub 2021 Oct 8. PMID 34625454
- [Background] McGirt MJ, Rossi V, Peters D, Dyer H, Coric D, Asher AL, Pfortmiller D, Adamson T. Anterior Cervical Discectomy and Fusion in the Outpatient Ambulatory Surgery Setting: Analysis of 2000 Consecutive Cases. Neurosurgery. 2020 Mar 1;86(3):E310-E315. doi: 10.1093/neuros/nyz514. PMID 31819994
- [Background] Garringer SM, Sasso RC. Safety of anterior cervical discectomy and fusion performed as outpatient surgery. J Spinal Disord Tech. 2010 Oct;23(7):439-43. doi: 10.1097/BSD.0b013e3181bd0419. PMID 20087224
- [Background] Arnold PM, Rice LR, Anderson KK, McMahon JK, Connelly LM, Norvell DC. Factors affecting hospital length of stay following anterior cervical discectomy and fusion. Evid Based Spine Care J. 2011 Aug;2(3):11-8. doi: 10.1055/s-0030-1267108. PMID 23532355
- [Background] Mariappan R, Mehta J, Massicotte E, Nagappa M, Manninen P, Venkatraghavan L. Effect of superficial cervical plexus block on postoperative quality of recovery after anterior cervical discectomy and fusion: a randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):883-90. doi: 10.1007/s12630-015-0382-3. Epub 2015 Apr 14. PMID 25869024
- [Background] Woldegerima YB, Hailekiros AG, Fitiwi GL. The analgesic efficacy of bilateral superficial cervical plexus block for thyroid surgery under general anesthesia: a prospective cohort study. BMC Res Notes. 2020 Jan 28;13(1):42. doi: 10.1186/s13104-020-4907-7. PMID 31992341
- [Background] Mulcahy MJ, Elalingam T, Jang K, D'Souza M, Tait M. Bilateral cervical plexus block for anterior cervical spine surgery: study protocol for a randomised placebo-controlled trial. Trials. 2021 Jun 29;22(1):424. doi: 10.1186/s13063-021-05377-4. PMID 34187541
- [Background] Hassan AH, Amer IA, Abdelkareem AM. Comparative study between dexmedetomidine versus dexamethasone as adjuvants to levobupivacaine for cervical plexus block in patients undergoing thyroid operation. prospective-randomized clinical trial. The Egyptian Journal of Hospital Medicine. 2021 Jul 1;84(1):1638-43.
- [Background] Al-Mustafa MM, Abu-Halaweh SA, Aloweidi AS, Murshidi MM, Ammari BA, Awwad ZM, Al-Edwan GM, Ramsay MA. Effect of dexmedetomidine added to spinal bupivacaine for urological procedures. Saudi Med J. 2009 Mar;30(3):365-70. PMID 19271064
- [Background] Vuyk J, Sitsen E, Reekers M. Intravenous Anesthetics. In: Miller RD, Eriksson LI, Cohen NH, Fleisher LA, Wiener-Kronish JP, Young WL, editors. Miller's Anesthesia. 8th ed. Philadelphia: Elsevier Churchill Livingstone; 2015. pp. 854-9
- [Background] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Background] Richard B, Alan JR, Vincent WS, Miller RD, Eriksson LI, Wiener-Kronish JP, Young WL. Spinal, epidural, and caudal anesthesia. Miller's anesthesia. 8th ed. Philadelphia, PA: Saunders, an imprint of Elsevier Inc. 2015:1684-720.
- [Background] Omar Mostafa M, Makram Botros J, Sayed Khaleel AM. Effect of Dexmedetomidine Versus Nalbuphine as an Adjuvant on Paravertebral Block to Manage Postoperative Pain After Mastectomies. Anesth Pain Med. 2018 Apr 28;8(2):e13308. doi: 10.5812/aapm.13308. eCollection 2018 Apr. PMID 30027066
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Chinnappa V, Chung F.What Criteria Should Be Used for Discharge after Outpatient Surgery?. InEvidence-Based Practice of Anesthesiology 2013 Jan 1 (pp. 343-351).
- [Background] Shi W, Dong J, Chen JF, Yu H. A meta-analysis showing the quantitative evidence base of perineural nalbuphine for wound pain from upper-limb orthopaedic trauma surgery. Int Wound J. 2023 May;20(5):1476-1490. doi: 10.1111/iwj.14002. Epub 2022 Nov 3. PMID 36330591